CLINICAL TRIAL: NCT02516501
Title: Investigating the Impact of a Ketogenic Diet Intervention During Radiotherapy on Body Composition: A Pilot Trial
Brief Title: Impact of a Ketogenic Diet Intervention During Radiotherapy on Body Composition
Acronym: KETOCOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MVZ Leopoldina GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15025
Record Dates: First submitted 2015-07-31; First posted 2015-08-06 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Neoplasms
Keywords: Ketogenic Diet; Body composition; Radiation therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Control group that will not receive advice to follow a ketogenic diet or reduce carbohydrates.
  Interventions: Radiation: Radio(chemo)therapy
- Intervention group 1 (Experimental): Patients who will receive each radiotherapy (RT) fraction after an overnight fast and subsequently ingest a ketogenic breakfast consisting of (i) up to 250 ml of a medium chain triglyceride drink (betaquik, vitaflo) plus (ii) 10g amino acids (MyAmino, dr. reinwald gmbh + co kg).
  Interventions: Dietary Supplement: MyAmino; Dietary Supplement: betaquik; Radiation: Radio(chemo)therapy
- Intervention group 2 (Experimental): Patients who will follow a ketogenic diet throughout the whole period of RT, Patients don't have to fast prior to each RT fraction, but will receive MyAmino analogous to Intervention group 1.
  Interventions: Dietary Supplement: MyAmino; Radiation: Radio(chemo)therapy

INTERVENTIONS:
Dietary Supplement: MyAmino — MyAmino is a supplement containing the eight essential amino acids. MyAmino has a theoretical net nitrogen utilization of 99%, so that almost no glucose will be created out of the maino acids.
  Other Names: Master amino acid pattern (MAP)
  Arms: Intervention group 1; Intervention group 2
Dietary Supplement: betaquik — betaquik is a medium chain triglyceride (MCT) emulsion. One bottle is 225ml corresponding to 45g MCT fats.
  Arms: Intervention group 1
Radiation: Radio(chemo)therapy — Radio(chemo)therapy as recommended by the institutional interdisciplinary tumor board.

SUMMARY:
Type of study: Pilot / phase I trial

Study purpose To assess the impact of a dietary intervention during radio(chemo)therapy (RCT) on body composition changes

Trial Treatment Patients will be split into a control group and intervention group 1. If willing to undertake a ketogenic diet for the duration of radiotherapy, patients are entered into intervention group 2.

* Group 1: On irradiation days irradiation after overnight fast + ketogenic breakfast consisting of 50-250 ml betaquik® (vitaflo, Bad Homburg, Germany) and 10g MyAmino (dr. reinwald healthcare gmbh + co kg, Altdorf, Germany).
* Group 2: Complete ketogenic diet plus 10g MyAmino/day
* Control: No dietary intervention.
* All groups: Weight measurements and bioimpedance analysis (BIA) once per week, routine blood parameters and quality of life (QoL) questionnaire before, during and after RCT

Endpoints

Primary:

* Feasibility of the dietary intervention during RCT, measured by dropout rates
* Changes in body weight
* BIA phase angle and quantities derived from BIA variables

Secondary:

* QoL
* Toxicities
* Blood parameters
* Grade of regression at time of surgery in case of rectum carcinomas

Inclusion criteria

* One of the following tumor entities:

  * Breast carcinoma
  * Rectum carcinoma
  * Head & Neck Cancer
* Histological confirmation of malignancy
* Signed written informed consent
* Karnofsky index ≥ 70
* Age between 18 and 75 years
* BMI between 18 and 34 kg/m^2

Exclusion criteria

* Palliative patients, in particular with metastasis
* Type I diabetes
* Pregnancy
* Pacemaker and other metallic parts within the body
* Known defects in enzymes necessary for ketogenesis, ketolysis, fatty acid oxidation or gluconeogenesis
* Unable to speak or understand German
* Cognitive impairments or psychological disorders
* Renal insufficiency

Planned accrual

* 15 patients with colorectal and mammary tumor plus 5 patients with H&N cancer in intervention group 1
* 15 patients with colorectal and mammary tumor plus 5 patients with H&N cancer in control group
* Minimum 5 patients of each tumor entity in intervantion group 2 Total: n ≥ 85 patients

Study procedure

1. Inclusion and full written informed consent.
2. Baseline BIA measurement and blood work
3. RCT with weekly BIA assessments; at least one blood withdrawal ± concurrent dietary intervention
4. Final BIA measurement and blood work after radiotherapy

Follow up For rectal carcinoma: Regression at time of surgery (c and p)

ELIGIBILITY:
Inclusion Criteria:

* RT of one of the following tumor entities: Mammary carcinoma, colorectal carcinoma, head and neck carcinoma
* Histologicallý confirmed malignant Tumor
* Written informed consent
* Karnofsky index >= 70
* 18 kg/m^2 < BMI < 34 kg/m^2

Exclusion Criteria:

* Palliative Treatment
* Type I Diabetes
* Pregnancy
* Pacemaker and othe rmetallic parts that make BIA predictions unreliable
* Unable to understand and speak German
* Cognitive impairments
* Renal insufficiency
* intake of carboanhydrase-inhibitors
* Rare metabolic disorders that speak against a ketogenic diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Dropout rate | 5-6 weeks
  Dropout rates (intervention groups 1+2) to assess feasibility/tolerability of the intervention
Body composition | 5-6 weeks
  This is a composite measure of several parameters obtained from the bioimpedance scale (mBCA 515, seca Germany). Body weight and composition derived from bioimpedance analysis will be assessed at least once per week. Body composition is composed of fat mass, fat free mass, total body water, extracellular water and intracellular water.
Phase angle | 5-6 weeks
  The phase angle is a raw parameter of bioimpedance analysis and will be tracked weekly at a total of 19 frequencies (1, 1.5,2,3,5,7.5,10,15,20,30,50,75,100,150,200,300,500,1000 kHz). The Focus will be on the Phase angle at 50kHz which is a standard frequency of most BIA devices.

SECONDARY OUTCOMES:
Quality of life | 5-6 weeks
  Evaluation of quality of life using EORTC QLQ-C30 and site-specific questionnaires at start, in the middle and at the end of RT.
Blood parameters | Blood parameters will be determined up to one week before the first RT fraction, at least once during their RT course (after an expected 3 weeks) and during their last week of RT..
  This is a composite measure of relevant blood parameters including small blood count, glucose, albumin, urea, HbA1c, beta-hydroxybutyrate, triglycerides, HDl and LDL cholesterol, creatinine, liver enzymes, insulin, IGF-1, TSH, free T3 and T4.
Regression grade (TNM classification) | 12 weeks
  Only for colorectal carcinoma patients undergoing neoadjuvant RT: cTN status prior to and ypTN status after surgery
Normal tissue toxicity after RT | 5-6 weeks
  Toxicity related to RT evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer J Klement, PhD, Principal Investigator — Department of Radiation Oncology, Leopoldina Hospital Schweinfurt
Locations (1):
- Department of Radiotherapy and Radiation Oncology, Schweinfurt, Bavaria, Germany

REFERENCES:
- [Background] Klement RJ, Sweeney RA. Impact of a ketogenic diet intervention during radiotherapy on body composition: I. Initial clinical experience with six prospectively studied patients. BMC Res Notes. 2016 Mar 5;9:143. doi: 10.1186/s13104-016-1959-9. PMID 26946138
- [Background] Klement RJ, Schafer G, Sweeney RA. A fatal case of Fournier's gangrene during neoadjuvant radiotherapy for rectal cancer. Strahlenther Onkol. 2019 May;195(5):441-446. doi: 10.1007/s00066-018-1401-4. Epub 2018 Nov 23. PMID 30470845
- [Background] Klement RJ, Sweeney RA. Impact of a ketogenic diet intervention during radiotherapy on body composition: II. Protocol of a randomised phase I study (KETOCOMP). Clin Nutr ESPEN. 2016 Apr;12:e1-e6. doi: 10.1016/j.clnesp.2015.11.001. Epub 2016 Jan 15. PMID 28531663
- [Result] Klement RJ, Schafer G, Sweeney RA. A ketogenic diet exerts beneficial effects on body composition of cancer patients during radiotherapy: An interim analysis of the KETOCOMP study. J Tradit Complement Med. 2019 Mar 21;10(3):180-187. doi: 10.1016/j.jtcme.2019.03.007. eCollection 2020 May. PMID 32670812
- [Result] Klement RJ, Champ CE, Kammerer U, Koebrunner PS, Krage K, Schafer G, Weigel M, Sweeney RA. Impact of a ketogenic diet intervention during radiotherapy on body composition: III-final results of the KETOCOMP study for breast cancer patients. Breast Cancer Res. 2020 Aug 20;22(1):94. doi: 10.1186/s13058-020-01331-5. PMID 32819413
- [Result] Klement RJ, Weigel MM, Sweeney RA. A ketogenic diet consumed during radiotherapy improves several aspects of quality of life and metabolic health in women with breast cancer. Clin Nutr. 2021 Jun;40(6):4267-4274. doi: 10.1016/j.clnu.2021.01.023. Epub 2021 Jan 27. PMID 33551218
- [Result] Klement RJ, Koebrunner PS, Meyer D, Kanzler S, Sweeney RA. Impact of a ketogenic diet intervention during radiotherapy on body composition: IV. Final results of the KETOCOMP study for rectal cancer patients. Clin Nutr. 2021 Jul;40(7):4674-4684. doi: 10.1016/j.clnu.2021.05.015. Epub 2021 May 31. PMID 34233255
- [Result] Klement RJ, Meyer D, Kanzler S, Sweeney RA. Ketogenic diets consumed during radio-chemotherapy have beneficial effects on quality of life and metabolic health in patients with rectal cancer. Eur J Nutr. 2022 Feb;61(1):69-84. doi: 10.1007/s00394-021-02615-y. Epub 2021 Jun 27. PMID 34175978
- [Result] Klement RJ, Sweeney RA. Impact of a ketogenic diet intervention during radiotherapy on body composition: V. Final results of the KETOCOMP study for head and neck cancer patients. Strahlenther Onkol. 2022 Nov;198(11):981-993. doi: 10.1007/s00066-022-01941-2. Epub 2022 May 2. PMID 35499696